CLINICAL TRIAL: NCT01264640
Title: The Impact of Aspirin and Clopidogrel on Brain-derived Neurotrophic Factor (BDNF) Concentrations in Human Serum and Plasma
Brief Title: Anti-Platelet Drugs and Brain-derived Neurotrophic Factor (BDNF) in Human Serum and Plasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Rostock (Other)
Responsible Party: PD Dr. Marek Lommatzsch, Abteilung für Pneumologie, University of Rostock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LO-0005
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-07

CONDITIONS: Healthy Volunteers
Keywords: Brain-derived neurotrophic factor (BDNF); Platelets; Aspirin; Clopidogrel
MeSH Terms: interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Intake of 500 mg Aspirin on day 1. Intake of 600 mg Clopidogrel on day 28. Measurement of platelet inhibition, platelet counts and BDNF, TGF-beta, 5-HT concentrations in peripheral blood on day 1 (before intake of 500 mg Aspirin), day 2 (24 hours after intake of 500 mg Aspirin), day 28 (before intake of 600 mg Clopidogrel), day 29 (24 hours after intake of 600 mg Clopidogrel).
  Interventions: Drug: Aspirin and Clopidogrel

INTERVENTIONS:
Drug: Aspirin and Clopidogrel — Intake of 500 mg Aspirin on day 1. Intake of 600 mg Clopidogrel on day 28. Blood collection for the measurement of platelet inhibition, platelet counts and BDNF, TGF-beta, 5-HT concentrations in peripheral blood on day 1 (before intake of 500 mg Aspirin), day 2 (24 hours after intake of 500 mg Aspirin), day 28 (before intake of 600 mg Clopidogrel), day 29 (24 hours after intake of 600 mg Clopidogrel).

SUMMARY:
The impact of anti-platelet drugs on the concentrations of Brain-derived neurotrophic factor (BDNF) in human plasma and serum is unknown. It is the aim of this study to investigate the impact of a single dose of Aspirin (500 mg) or Clopdigrel (600 mg) on the concentrations of Brain-derived neurotrophic factor (BDNF) in plasma and serum of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Gender: Male

Exclusion Criteria:

* Any acute disease
* Any chronic disease
* Any medication
* Allergies / Intolerance in association with Aspirin or Clopidogrel

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-02 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
BDNF plasma and serum concentration 24 hours after Aspirin or Clopidgrel intake | 24 hours

SECONDARY OUTCOMES:
5-HT and TGF-beta concentrations 24 hours after Aspirin or Clopidgrel intake | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marek Lommatzsch, PD Dr., Principal Investigator — University of Rostock
Locations (1):
- Dep. of Pneumology, University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Lommatzsch M, Zingler D, Schuhbaeck K, Schloetcke K, Zingler C, Schuff-Werner P, Virchow JC. The impact of age, weight and gender on BDNF levels in human platelets and plasma. Neurobiol Aging. 2005 Jan;26(1):115-23. doi: 10.1016/j.neurobiolaging.2004.03.002. PMID 15585351
- See also: Website of the Medical faculty of the University of Rostock — http://www.med.uni-rostock.de